CLINICAL TRIAL: NCT05853978
Title: The Evaluation of Balanced Salt Solution During Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adam Fedyk, MD, FACS (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Adam Fedyk, MD, FACS, Owner, St. Louis Eye Institute
Organization: St. Louis Eye Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ARF-23-001
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Fuchs Dystrophy; Cataract
Keywords: Fuchs Corneal Endothelial Dystrophy; Nuclear Sclerosis; Cataract Surgery; Paired Eye; ARF-23-001
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract | interventions — glutathione-bicarbonate-Ringer solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BSS Plus (Experimental)
  Interventions: Drug: BSS Plus
- BSS (Active Comparator)
  Interventions: Drug: BSS

INTERVENTIONS:
Drug: BSS Plus — BSS PLUS® Sterile Intraocular Irrigating Solution (balanced salt solution enriched with bicarbonate, dextrose, and glutathione)
  Arms: BSS Plus
Drug: BSS — BSS® Sterile Irrigating Solution (balanced salt solution)
  Arms: BSS

SUMMARY:
This study aims to identify if the use of BSS PLUS® Sterile Intraocular Irrigating Solution as an irrigation solution leads to improved corneal outcomes vs BSS® Sterile Irrigating Solution in more compromised corneas.

ELIGIBILITY:
Inclusion Criteria

1. Adults, 22 years of age or older, with bilateral visually significant cataracts.
2. Subjects with Fuch's Dystrophy that present with:

   1. nonconfluent and confluent guttata; and/or
   2. CCT > 580 microns.
3. Unremarkable systemic health but inclusive of controlled type II diabetes and hypertension
4. Ability to comprehend and sign a statement of informed consent.
5. Ability to complete all required postoperative visits.
6. Willingness to use at least one medically acceptable form of birth control throughout the duration of study participation. (for female subjects of childbearing potential only).

Exclusion Criteria

1. Planned implantation of multifocal intraocular lenses.
2. Planned secondary procedure(s) to occur in conjunction with cataract surgery (i.e., goniotomy)
3. History of severe dry eye.
4. Retinal and retinal vascular pathologies, age-related macular degeneration
5. Uncontrolled systematic diseases, including: hypertension, diabetes, systemic cardiovascular diseases and hematological diseases.
6. Autoimmune disease such as rheumatoid arthritis.
7. Female subjects of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Central Corneal Thickness (CCT) | Postoperative: Day 1
  Changes in central corneal thickness following cataract surgery with BSS PLUS® Sterile Intraocular Irrigating Solution, as compared to BSS® Sterile Irrigating Solution

SECONDARY OUTCOMES:
Intraoperative Grading of Corneal Edema | Day 0
  Intraoperative grading of corneal edema during cataract surgery with BSS PLUS® Sterile Intraocular Irrigating Solution, as compared to BSS® Sterile Irrigating Solution.
Number of Intraocular Irrigating Solution Drops Used | Day 0
  Number of BSS PLUS® Sterile Intraocular Irrigating Solution drops used during cataract surgery to rewet corneal surface and maintain clarity, as compared to BSS® Sterile Irrigating Solution.

OTHER OUTCOMES:
Corneal Surface Keratopathy and Conjunctival Staining | Postoperative: Day 1 and Week 1
  Changes in corneal surface keratopathy and conjunctival staining following cataract surgery with BSS PLUS® Sterile Intraocular Irrigating Solution, as compared to BSS® Sterile Irrigating Solution.
Conjunctival Injection | Postoperative: Day 1 and Week 1
  Changes in conjunctival injection following cataract surgery with BSS PLUS® Sterile Intraocular Irrigating Solution, as compared to BSS® Sterile Irrigating Solution.
Ocular Comfort Index (OCI) | Postoperative: Day 1 and Week 1
  Assessment of Ocular Comfort Index (OCI) following cataract surgery with BSS PLUS® Sterile Intraocular Irrigating Solution, as compared to BSS® Sterile Irrigating Solution.
Best Corrected Visual Acuity (BCVA) | Postoperative: Month 1
  Best Corrected Visual Acuity (BCVA) following cataract surgery with BSS PLUS® Sterile Intraocular Irrigating Solution, as compared to BSS® Sterile Irrigating Solution.
Endothelial Cell Density (ECD) | Postoperative: Month 1
  Endothelial Cell Density (ECD) following cataract surgery with BSS PLUS® Sterile Intraocular Irrigating Solution, as compared to BSS® Sterile Irrigating Solution.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Louis Eye Institute, Town and Country, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided